CLINICAL TRIAL: NCT06901596
Title: Sugammadex Reduces Antiemetic Effect of Dexamethasone
Status: Not yet recruiting | Type: Observational
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Efrain Riveros Perez, MD, Associate Professor of Anesthesiology, Augusta University
Other Study IDs: 2204574
Record Dates: First submitted 2025-03-19; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: PONV
Keywords: sugammadex; dexamethasone; PONV; perioperative; surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dexamethasone: Surgical patients who received dexamethasone as prophylactic antiemetic
- Dexamethasone + sugammadex: Patients who received dexamethasone intraoperatively and sugammadex to reverse muscle relaxation

SUMMARY:
Sugammadex is a medication used for reversal of muscle relaxation during procedures under general anesthesia. It works by encapsulating muscle relaxant molecules with a steroid ring in its structure. On the other hand, postoporative nause and vomiting (PONV) is an adverse outcome during anesthesia. PONV can be prevented with pharmacologic agents such as ondansetron and dexamethasone. Dexamethasone is a steroidal agent that can interact with sugammadex. In theory, this interaction could lead to reduced effectiveness of sugammadex. In fact, several studies have explored this interaction. However, the effect of sugammadex on the antiemetic effect of dexamethasone has not been evaluated. This study intends to evaluate this interaction.

DETAILED DESCRIPTION:
The study will use de-identified retrospective data to conduct a cross-sectional study to determine the effect of sugammadex on the antiemetic efficacy of dexamethasone in elective adult surgical patients who underwent surgery in a tertiary care center between January 1 2023 and January 1 2024 . The investigators will conduct univariate and multivariate analysis to assess the effect.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* Elective surgery
* ASA 1, 2, 3
* At least one risk factor for PONV

Exclusion Criteria:

* Pregnancy
* Receiving antiemetics prior to arrival to preoperative holding area
* Receiving opioids prior to arrival to preoperative holding area
* Admission to ICU
* Altered mental status
* Rapid sequence induction
* Nausea or vomiting before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult surgical patients scheduled for elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Rate of PONV | 2 hours after admission to PACU
  Number of events of PONV during 2 hours after admission to PACU

IPD SHARING:
Plan to Share IPD: No
Data are de-identified. The data used for data analysis can be available upon request

REFERENCES:
- [Background] Park HY, Choi HR, Kim YB, Oh SK, Kim T, Yang HS, In J. Chronic exposure to dexamethasone may not affect sugammadex reversal of rocuronium-induced neuromuscular blockade: an in vivo study on rats. Anesth Pain Med (Seoul). 2023 Jul;18(3):275-283. doi: 10.17085/apm.23021. Epub 2023 Jul 14. PMID 37468197
- [Background] Choi H, Park SY, Kim YB, In J, Yang HS, Lee JS, Kim S, Park S. Effects of dexamethasone and hydrocortisone on rocuroniuminduced neuromuscular blockade and reversal by sugammadex in phrenic nerve-hemidiaphragm rat model. Korean J Anesthesiol. 2019 Aug;72(4):366-374. doi: 10.4097/kja.d.18.00238. Epub 2019 Mar 19. PMID 30886132
- [Background] Koo CH, Hwang JY, Min SW, Ryu JH. A Meta-Analysis on the Effect of Dexamethasone on the Sugammadex Reversal of Rocuronium-Induced Neuromuscular Block. J Clin Med. 2020 Apr 24;9(4):1240. doi: 10.3390/jcm9041240. PMID 32344687
- [Background] Lim BG, Won YJ, Kim H. The effect of dexamethasone on sugammadex reversal of rocuronium-induced neuromuscular blockade in surgical patients undergoing general anesthesia: A systematic review and meta-analysis. Medicine (Baltimore). 2021 Feb 5;100(5):e23992. doi: 10.1097/MD.0000000000023992. PMID 33592855
- [Background] Batistaki C, Pandazi A, Kyttari A, Kaminiotis E, Kostopanagiotou G. Is there an interaction between dexamethasone and sugammadex in real clinical conditions? A randomized controlled trial in patients undergoing laparoscopic cholecystectomy. J Anaesthesiol Clin Pharmacol. 2019 Apr-Jun;35(2):215-219. doi: 10.4103/joacp.JOACP_42_17. PMID 31303711